CLINICAL TRIAL: NCT03549845
Title: Pragmatic Randomized Controlled Trial of the Cardiovascular Health Awareness Program (CHAP) in Subsidized Social Housing
Brief Title: Cardiovascular Health Awareness Program (CHAP) in Subsidized Social Housing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Université de Montréal (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CHAP052018
Record Dates: First submitted 2018-05-15; First posted 2018-06-08 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Cardiovascular Diseases; Cardiovascular Risk Factor; Diabetes Mellitus
Keywords: Healthcare Utilization; Emergency Department; Hospitalization; Low Income; Social Housing; Older Adults; Quality of Life
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Emergencies

STUDY DESIGN:
Intervention Model Description: Pragmatic cluster randomized controlled trial with parallel intervention and control groups.
  Randomization will occur at the building level (clusters) and the intervention is open to all building residents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHAP Intervention (Experimental): The Cardiovascular Health Awareness Program (CHAP) intervention is an on-site drop-in, monthly, cardiovascular risk assessment program run by trained volunteers with community-led group health sessions that deliver education and information about access to community health resources. The education sessions will be delivered by national and provincial and local community organizations utilizing already developed material as much as possible, but maintaining consistency across both provinces. Health education sessions will include topics such as: Physical Activity, Healthy Eating, Stress, Tobacco Use, High Blood Pressure, Role of Pharmacist: How they can assist people, and Appropriate use of 9-1-1. This intervention will be held in a common room in selected subsidized housing buildings.
  Interventions: Behavioral: Cardiovascular Health Awareness Program
- Control (No Intervention): The control buildings will receive usual care which will be wellness programs already present in the building prior to the RCT if these are present. Not all control buildings will have wellness programs.

INTERVENTIONS:
Behavioral: Cardiovascular Health Awareness Program — Cardiovascular disease prevention and health promotion
  Arms: CHAP Intervention

SUMMARY:
This project aims to improve the cardiovascular health of seniors living in subsidized housing by implementing the successful community-based Cardiovascular Health Awareness Program (CHAP). CHAP is a patient-centred, interdisciplinary, multi-pronged, community-led CVD and stroke prevention and management program designed to prevent and reduce the impact of cardiovascular disease in older adults. The program addresses common cardiovascular disease risk factors, such as smoking, physical activity and poor diet by raising awareness of health and community resources available to encourage self-care and appropriate management of cardiovascular disease. A randomized controlled trial will be used to evaluate the impact of CHAP on healthcare utilization by older adults living in subsidized housing.

DETAILED DESCRIPTION:
This project aims to improve the cardiovascular health of seniors living in subsidized housing by implementing the successful community-based Cardiovascular Health Awareness Program (CHAP). Residents in subsidized housing are considered to be a vulnerable population because of their low income and tend to be in poorer health; with a multitude of chronic illnesses, such as cardiovascular disease (CVD) and diabetes.

This project will build on the success of CHAP in other provinces. The program has been shown to reduce blood pressure and CVD-related hospitalization costs. CHAP is a patient-centred, interdisciplinary, multi-pronged, community-led CVD and stroke prevention and management program designed to prevent and reduce the impact of cardiovascular disease in older adults. The program addresses common cardiovascular disease risk factors, such as smoking, physical activity and poor diet by raising awareness of health and community resources available to encourage self-care and appropriate management of cardiovascular disease.

Taking the form of a randomized controlled trial, the sample will be subsidized housing buildings (low income) for those aged 55 years and over. During CHAP monthly assessment sessions, participants will 1) complete a consent form, 2) complete a cardiovascular risk profile form, 3) undergo blood pressure measurement using an automated blood pressure measuring device, 4) receive targeted healthy lifestyle and preventive care materials, 5) be invited to participate in group health education sessions. Those patients identified at high risk will be assessed by a health professional and referred to a family physician for timely and appropriate follow-up.. The impact this program will have on health care utilization (emergency visits, cardiovascular hospitalization rates) will be measured using administrative databases.

ELIGIBILITY:
Building Inclusion Criteria:

* Approximately 50-200 apartment units
* Majority of residents are 55 years of age or older.
* Unique postal code
* Availability of at least one building with similar characteristics for matching/randomization

Individual Inclusion Criteria

* Resides in a study building
* Aged 55 years or older
* Speaks and reads English or French

Note: Younger residents will be allowed to take part in the program but their data will not be included in the analysis.

Exclusion Criteria:

* None

Min Age: 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2742 (Actual)
Dates: Start 2018-09-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Healthcare Utilization Composite - Change in CVD-related emergency department visits and hospitalizations | Monthly from 1 year pre-intervention to 1 year post-intervention
  Change in rate of CVD-related emergency department visits and hospitalizations by postal code from administrative databases (Building-level analysis)

SECONDARY OUTCOMES:
Healthcare Utilization - Change in all-cause emergency department visits | Monthly from 1 year pre-intervention to 1 year post-intervention
  Change in rate of all-cause emergency department visits by postal code from administrative
Healthcare Utilization - Change in all-cause hospitalizations | Monthly from 1 year pre-intervention to 1 year post-intervention
  Change in all-cause hospitalization rates by postal code from administrative data (building-level)
Change in quality of life | Baseline and 1 year
  Measured using EQ-5D-5L
Quality-Adjusted Life Years (QALYs) | 1 year (post-intervention)
  Calculated from EQ-5D-5L at two time points and Canadian value sets
Cost-effectiveness | 1 year (post-intervention)
  Calculated from program cost data and health outcomes
Participant experience of the CHAP intervention | 1 year (post-intervention)
  Participant experience of the intervention will be evaluated through qualitative individual interviews and focus groups of residents.

OTHER OUTCOMES:
Cardiovascular Risk - Change in blood pressure | Baseline and 1 year
  Change in measured blood pressure (automated, validated device)
Cardiovascular Risk - Change in body mass index | Baseline and 1 year
  Change in body mass index calculated from height and weight (self-reported)
Cardiovascular Risk - Change in waist circumference | Baseline and 1 year
  Change in waist circumference (measured with measuring tape)
Cardiovascular Risk - Change in diabetes risk score | Baseline and 1 year
  Change in diabetes risk score (CANRISK questionnaire)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Agarwal, Principal Investigator — McMaster University; Janusz Kaczorowski, Principal Investigator — CHUM (Université de Montréal)
Locations (1):
- Centre de recherche du CHUM, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
There is currently no plan for individual participant data to be shared. Aggregate data will be shared upon request.

REFERENCES:
- [Derived] Agarwal G, Girard M, Angeles R, Pirrie M, Lussier MT, Marzanek F, Dolovich L, Paterson JM, Thabane L, Kaczorowski J. Design and rationale for a pragmatic cluster randomized trial of the Cardiovascular Health Awareness Program (CHAP) for social housing residents in Ontario and Quebec, Canada. Trials. 2019 Dec 23;20(1):760. doi: 10.1186/s13063-019-3806-5. PMID 31870415